CLINICAL TRIAL: NCT02479074
Title: The Utility of feNO in the Differential Diagnosis of Chronic Cough: The Response to Anti-inflammatory Therapy With Prednisolone and Montelukast
Brief Title: The Utility of feNO in the Differential Diagnosis of Chronic Cough
Acronym: TUF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: Aerocrine AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: AcadMed1002015
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cough
Keywords: Chronic
MeSH Terms: conditions — Cough; Bronchiolitis Obliterans Syndrome | interventions — montelukast; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Montelukast (high FeNO) (Active Comparator): Montelukast 10 mg film-coated tablet contains montelukast sodium equivalent to 10 mg montelukast patients to take one tablet per day for 28 days Montelukast is a Class B medicine
  Interventions: Drug: Montelukast (High FeNO group)
- Prednisolone, Montelukast (high FeNO) (Active Comparator): Prednisolone 5 mg and montelukast 10 mg. Patients to take Prednisolone 5 mg, 4 tablets per day for 14 days patients to take Montelukast 10 mg film-coated tablet per day for another 14 days Prednisolone is a Class A medicine Montelukast is a Class B medicine
  Interventions: Drug: Prednisolon, Montelukast (High FeNO)
- Montelukast (Active Comparator): Montelukast 10 mg film-coated tablet contains montelukast sodium equivalent to 10 mg montelukast patients to take one tablet per day for 28 days Montelukast is a Class B medicine
  Interventions: Drug: Montelukast (Low FeNO group)

INTERVENTIONS:
Drug: Montelukast (High FeNO group) — Montelukast 10 mg film-coated tablet contains montelukast sodium equivalent to 10 mg montelukast patients to take (oral use) one tablet per day for 28 days
  Other Names: Montelukast
  Arms: Montelukast (high FeNO)
Drug: Prednisolon, Montelukast (High FeNO) — Prednisolone 5 mg, patients to take 4 tablets per day for 14 days then take Montelukast 10 mg tablet per day for another 14 days.
  Other Names: Prednisolone and Montelukast
  Arms: Prednisolone, Montelukast (high FeNO)
Drug: Montelukast (Low FeNO group) — Montelukast 10 mg film-coated tablet contains montelukast sodium equivalent to 10 mg montelukast patients to take one tablet per day for 28 days
  Other Names: Montelukast
  Arms: Montelukast

SUMMARY:
In this study the investigators wish to explore the difference in 24 hr. cough counts measured using the Hull Automated Cough Counter (HACC), from baseline and after two weeks treatment with either montelukast or prednisolone in patients with an NO measurement of ≥30 ppb at screening.

DETAILED DESCRIPTION:
Patients attending the unit as part of their normal outpatients' appointment will be approached with regards to whether interested in taking part in the study. During an outpatients appointment all new chronic cough patients undertake Demographics assessment, full blood count, spirometry test, FeNO measurement and concomitant medication as part of their standard medical care. If a patient decides to take part in this study then at this visit they will have further tests outside their standard medical care including, sputum induction, completion of Leicester cough questionnaire, cough challenge and 24 hr cough monitoring at the screening visit. All the data collected in terms of the clinic visit and additional tests will be analysed in this study.

40 patients with chronic cough and a FeNO≥30 ppb will be enrolled in to the High FeNO Treatment Groups. They will be randomised on a 1:1 ratio to receive either: Montelukast 10 mg daily for four weeks or Prednisolone 20 mg daily for two weeks followed by two weeks Montelukast 10 mg. 20 subjects with chronic cough and a FeNO≤20 ppb will be enrolled in low FeNO Treatment Group will receive montelukast 10 mg for 28 days.

The study consists of five visits to the unit. The first visit will be combined with the patients scheduled clinic appointment. During this visit the investigators will carry out some preliminary assessments such as checking medical history, physical examination, full blood count and vital signs. Demographics assessments, spirometry test, FeNO measurement and concomitant medication will be recorded as per their scheduled clinic visit.

Further testing will be conducted with regards to the study, these tests include: sputum induction, cough challenge, Hull Airways Reflux Questionnaire (HARQ), Leicester Cough Questionnaire (LCQ) and 24h cough monitoring all these tests will be operated at baseline and after 2 weeks and 4 weeks treatment.

Also pregnancy test for women of child bearing potential is required in this study.

At the end of visit 1, patients will receive 14 or 28 days' supply of the randomised study medication.

Visit 2 (13th day) and visit 4 (27th day): Participants will be asked to come to the unit where The Hull Automated Cough Counter will be applied to measure their cough frequency for 24 hours at the end of their treatment.

Visit 3 (14th day) and visit 5 (28th day): Patients will be assessed for any adverse events and any changes in concomitant medication use during the trial and also their vital signs will be checked. After that the FeNo measurement, Pulmonary Function Tests, cough challenge, sputum induction, 24h cough monitoring, Hull Airways Reflux Questionnaire (HARQ) and Leicester Cough Questionnaire (LCQ) will be repeated to compare with the first assessment.

At the end of the study all patients will be reviewed by a chronic cough registrar/consultant as per the standard care as a clinic patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic cough (at least 8 weeks duration)
* Male and female subjects of at least 18 yrs of age
* Subjects able to understand the study and co-operate with the study procedures
* Subjects who consent to their general practitioner (GP) being informed of their study participation.
* Patients with a FeNO of ≥30ppb at presentation to the Chronic cough clinic.( required for entry on to the high FeNO treatment groups)
* Patients with FeNO ≤ 20 ppb at presentation to the chronic cough clinic (required for entry as low FeNO treatment group)

Exclusion Criteria:

* Patients with current diagnosis of asthma.
* Female subjects who are pregnant, or lactating, or who are of child bearing potential but are not using contraceptive measures.
* Suffering from any concomitant disease (chronic heart, chronic lung such as; COPD, bronchiectasis and cystic fibrosis, chronic renal, chronic liver or neuromuscular disease or immunosuppression; pneumonia and diabetes) which may interfere with study procedures or evaluation.
* A lower respiratory tract infection 4 weeks prior to entry on to study
* Systemic infections
* Live virus immunisation planned within next 3 months
* Subjects with no previous chickenpox who had a recent (<=28 days) close personal contact with chickenpox OR herpes zoster (high FeNO treatment groups only)
* Subjects having recent (<=28 days) exposure to measles (high FeNO treatment groups only)
* Participation in another study (use of investigational product) within 30 days preceding entry on to study.
* Alcohol or drug abuse
* Inability to follow study procedures
* Use of corticosteroids either as inhaled, topical or systemic ≥ 4weeks prior to enrolment
* Subjects with known allergy to prednisolone, montelukast
* Subjects who are taking Angiotensin Converting Enzymes (ACE) inhibitors.
* Current smoker
* Subjects who are taking bronchodilators should be on it for at least 4 weeks on regular dose and carry on the same dose during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Hull Automated Cough counter | 28 days
  To determine the difference in objective measure of cough as demonstrated by 24 hr cough counts at the baseline, after 2 and 4 weeks treatment between three treatment groups with an associated elevated FeNO.

SECONDARY OUTCOMES:
HARQ and LCQ questionnaires | 28 days
  Compare change in subjective measures on HARQ and LCQ questionnaires of cough between the treatment groups at the baseline and after 2 week and 4 weeks treatment.
FVC as measured through spirometry | 28 days
  Compare change in FVC between treatment groups at the baseline and after 2 weeks and 4 weeks treatment.
Cough Challenge | 28 days
  Change in cough reflex sensitivity using inhaled citric acid between treatment groups at the baseline and after 2 weeks and 4 weeks treatment.
Sputum Induction | 28 days
  Change in Sputum inflammatory markers between treatment groups at the baseline and after 2 weeks and 4 weeks treatment.
Blood Count | Baseline
  Assess whether previous history of blood eosinophils may predict therapeutic response to anti-inflammatory medication in cough.
FeNO measurement | 28 days
  Assess whether the efficiency of FeNO may help to predict therapeutic response to anti-inflammatory medication in cough.

CONTACTS AND LOCATIONS:
Overall Officials: Alyn Morice, Professor, Principal Investigator — Head of Centre for Cardiovascular and Metabolic Studies
Locations (1):
- Respiratory Medicine, Clinical trials Unit, Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Background] Everett CF, Kastelik JA, Thompson RH, Morice AH. Chronic persistent cough in the community: a questionnaire survey. Cough. 2007 Mar 23;3:5. doi: 10.1186/1745-9974-3-5. PMID 17381836
- [Background] Ford AC, Forman D, Moayyedi P, Morice AH. Cough in the community: a cross sectional survey and the relationship to gastrointestinal symptoms. Thorax. 2006 Nov;61(11):975-9. doi: 10.1136/thx.2006.060087. Epub 2006 Jun 29. PMID 16809412
- [Background] Brightling CE, Ward R, Goh KL, Wardlaw AJ, Pavord ID. Eosinophilic bronchitis is an important cause of chronic cough. Am J Respir Crit Care Med. 1999 Aug;160(2):406-10. doi: 10.1164/ajrccm.160.2.9810100. PMID 10430705
- [Background] Korevaar DA, Westerhof GA, Wang J, Cohen JF, Spijker R, Sterk PJ, Bel EH, Bossuyt PM. Diagnostic accuracy of minimally invasive markers for detection of airway eosinophilia in asthma: a systematic review and meta-analysis. Lancet Respir Med. 2015 Apr;3(4):290-300. doi: 10.1016/S2213-2600(15)00050-8. Epub 2015 Mar 20. PMID 25801413
- [Background] Sadeghi MH, Wright CE, Hart S, Crooks M, Morice AH. Does FeNO Predict Clinical Characteristics in Chronic Cough? Lung. 2018 Feb;196(1):59-64. doi: 10.1007/s00408-017-0074-6. Epub 2017 Nov 25. PMID 29177539
- [Result] Dicpinigaitis PV, Dobkin JB, Reichel J. Antitussive effect of the leukotriene receptor antagonist zafirlukast in subjects with cough-variant asthma. J Asthma. 2002 Jun;39(4):291-7. doi: 10.1081/jas-120002285. PMID 12095178
- [Derived] Sadeghi MH, Wright CE, Hart S, Crooks M, Morice A. Phenotyping patients with chronic cough: Evaluating the ability to predict the response to anti-inflammatory therapy. Ann Allergy Asthma Immunol. 2018 Mar;120(3):285-291. doi: 10.1016/j.anai.2017.12.004. PMID 29508715